CLINICAL TRIAL: NCT00693134
Title: The Role of Matrix Metalloproteinases and Tissue Inhibitors of Metalloproteinases in Children With Acute Inflammatory Cardiomyopathy
Brief Title: Role of Matrix Metalloproteinases (MMPs) and Tissue Inhibitors of Metalloproteinases (TIMPs) in Children With Myocarditis
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Tia Tortoriello-Raymond, MD, Universtty of Texas - Southwestern Medical Center
Other Study IDs: 012004-072
Record Dates: First submitted 2008-06-04; First posted 2008-06-06 (Estimated); Last update posted 2008-06-06 (Estimated); Status verified 2008-02

CONDITIONS: Myocarditis
MeSH Terms: conditions — Myocarditis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biopsy tissue, if available.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Myocarditis Patients: Patients initially diagnosed with myocarditis.
- Control Patients: Patients with no known cardiomyopathies

SUMMARY:
Children can have or develop certain problems with their heart function, specifically with the heart muscle or myocardium. This problem can be caused by many things specifically by infection resulting in myocarditis (inflammation of the heart muscle) or dilated cardiomyopathy (caused by many factors including high blood pressure and heart attacks). The body goes through many processes to repair the injured tissue including using proteins that cause the muscle mass to increase called matrix metalloproteinases (MMPs). The body also uses proteins that direct the MMPs to stop increasing the muscle mass called tissue inhibitory of metalloproteinases (TIMPs). Currently, there are no published studies that explain or evaluate the relationship that MMPs and TIMPs have in myocarditis and dilated cardiomyopathy in children.

The investigator wishes to perform a prospective study of the serum levels of these proteins and their regulators in children with myocarditis and/or dilated cardiomyopathy and compare them with children that have no heart disease.

DETAILED DESCRIPTION:
All children who present with signs and symptoms of myocarditis and have laboratory findings consistent with cardiomyopathy will be eligible. After prospective consent, all subjects will receive: (1) a complete physical examination, (2) complete transthoracic echocardiogram to better characterize the disease process. Follow-up echocardiograms will be performed at 24-72 hours after admission into the protocol and at discharge from the hospital. Approximately 2 teaspoons of blood will be drawn at: (1) enrollment, (2) 24 hours after, (3) 72 hours after, (4) and at hospital discharge. Those subjects that receive a heart transplant will have blood drawn at the time of transplantation. For those that have a cardiac catheterization or have a muscle biopsy as part of their standard of care, will also have a biopsy of their right ventricle performed.

Data to be collected: Minimum patient demographic data (age, sex, ethnic origin), vital signs, clinical course events/data (i.e. need for dialysis, length of stay, surgical time points, etc), diagnostic test results (EKGs, ECHOs, etc), significant medical history data, and standard of care laboratory results.

The investigator wishes to evaluate the relationship of this data with the patient's diagnosis, clinical course, and serum levels of MMP and TIMP proteinases.

ELIGIBILITY:
Inclusion Criteria:

1. Evidence from diagnostic tests and physical exam that confirm inflammatory cardiomyopathy.

Exclusion Criteria:

1. Patients with structural heart disease other than septal defects or patent ductus arteriosus
2. Patients with history of arrhythmia
3. Patients with history of ventricular dysfunction diagnosed by echocardiograms
4. Patients with history of chronic systemic illness

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Inpatients of the Cardiac Service at Children's Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2004-03; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Determine correlation between proteinases (MMPs and TIMPs) and their regulators in children with acute inflammatory cardiomyopathy. | Length of hospital stay from time of admission to protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Tia A Tortoriello-Raymond, MD, Principal Investigator — University of Texas - Southwestern Medical Center, Children's Medical Center
Locations (1):
- Children's Medical Center, Dallas, Texas, United States